CLINICAL TRIAL: NCT03067818
Title: Mechanisms of Arm Recovery in Stroke Patients With Hand Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: MedStar National Rehabilitation Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21HD090516-01 (NIH)
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Stroke; Hemiparesis; Cerebral Vascular Accident; Stroke, Ischemic
Keywords: arm; rehabilitation; non-invasive brain stimulation; transcranial magnetic stimulation; upper extremity
MeSH Terms: conditions — Stroke; Paresis; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Each participant will receive stimulation targeting each brain area. The order in which the stimulation sites are targeted for each participant is randomized and there is a washout period of several weeks between each treatment.
Who Masked: Outcomes Assessor
Masking Description: The individual that conducts the tests of arm movement will be unaware of which brain area was stimulated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unaffected Hemisphere (Experimental): Application of "Unaffected Transcranial Magnetic Stimulation" to unaffected hemisphere site prior to physical practice
  Interventions: Procedure: Unaffected Transcranial Magnetic Stimulation
- Affected Hemisphere (Experimental): Application of "Affected Transcranial Magnetic Stimulation" to affected hemisphere site prior to physical practice
  Interventions: Procedure: Affected Transcranial Magnetic Stimulation
- Control Site (Active Comparator): Application of "Control Transcranial Magnetic Stimulation" to control site prior to practice
  Interventions: Procedure: Control Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Unaffected Transcranial Magnetic Stimulation — Non-invasive brain stimulation to unaffected hemisphere site prior to practice
  Arms: Unaffected Hemisphere
Procedure: Affected Transcranial Magnetic Stimulation — Non-invasive brain stimulation to affected hemisphere site prior to practice
  Arms: Affected Hemisphere
Procedure: Control Transcranial Magnetic Stimulation — Non-invasive brain stimulation to control site prior to practice
  Arms: Control Site

SUMMARY:
This study examines the effect of non-invasive brain stimulation targeting different brain areas on movement of the affected arm post-stroke. Participants will receive stimulation to each of 3 different brain areas combined with a session of arm exercise.

DETAILED DESCRIPTION:
Small improvements in affected arm movement can be made with intensive physical practice. These improvements could potentially be enhanced by combining non-invasive brain stimulation with practice.

To develop such an intervention, it is necessary to understand which brain areas should be stimulated in which types of patients. It is probably more beneficial to target one side of the brain vs. the other, for example, depending on the characteristics of the stroke.

This study will examine the effect of stimulating one side of the brain vs. the other on the amount of improvement that occurs from physically practicing functional arm movements.

ELIGIBILITY:
Inclusion Criteria:

* More than 6 months post-stroke
* Loss of voluntary finger movement in the affected hand
* Some voluntary movement of affected shoulder and/or elbow

Exclusion Criteria:

* Brainstem or cerebellar stroke
* Severe cognitive or language deficits
* Epilepsy or other seizure disorder
* Central nervous system disease or disorder other than stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Change in movement time | Baseline and 1 Day
  Percentage change in time it takes to move the arm a standardized distance

SECONDARY OUTCOMES:
Change in maximum reaching distance | Baseline and 1 Day
  Percentage change in maximum distance participant is able to reach
Change in hand path kinematics | Baseline and 1 Day
  Percentage change in temporal and spatial movement of the hand during reaching

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Harris-Love, PhD, Principal Investigator — George Mason University
Locations (1):
- MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No